CLINICAL TRIAL: NCT06765096
Title: Impact of Virtual Reality Model for Pelvic Floor Anatomy on Users' Educational Level and Experience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/005397
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (VR) model for pelvic floor anatomy (Experimental): Participants will receive one session on educational virtual reality (VR) model for pelvic floor anatomy.
  Interventions: Other: Educational Virtual Reality Model

INTERVENTIONS:
Other: Educational Virtual Reality Model — Participants will receive one session on educational virtual reality (VR) model for pelvic floor anatomy.

SUMMARY:
The purpose of the study is to evaluate the impact of virtual reality (VR) model for pelvic floor anatomy on users' educational level and experience.

DETAILED DESCRIPTION:
Virtual reality (VR) has gained significant attention as an educational tool in various fields, including science and health education. Its capacity to create immersive, interactive environments allows students to explore complex, three-dimensional structures, enhancing visualization and understanding of abstract or intricate concepts. VR can bridge gaps in traditional education by offering experiences that are otherwise challenging to replicate in conventional classroom settings, such as real-time manipulation of anatomical models.

In health sciences, VR is particularly valuable for anatomy education. Studies have shown that VR's interactive and immersive nature fosters deeper comprehension, especially in understanding spatial relationships within anatomical structures. A VR model for pelvic floor anatomy could therefore serve as a powerful tool, allowing users to engage in a hands-on learning experience that enhances knowledge retention and user satisfaction.

Research indicates that VR may improve educational outcomes not only through knowledge acquisition but also by stimulating students' motivation and positive attitudes toward learning. A recent study has found that VR helped students develop problem-solving and visualization skills, which are crucial for disciplines requiring spatial awareness, such as anatomy. However, while VR shows promise, questions remain about its effectiveness compared to traditional educational methods, especially in specialized fields like pelvic floor anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Physical therapy undergraduate, graduate, and postgraduate students, as well as professionals.
* Participants must be physically able to wear and interact with a VR headset

Exclusion Criteria:

* Lack of Anatomy Background.
* Prior Extensive VR Experience in Anatomy.
* Severe Motion Sickness or Visual Disorders.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
A self-structured questionnaire | 1 month
  A self-structured questionnaire will serve as the primary data collection tool. The questionnaire is divided into eight sections, covering:
  * Demographics.
  * Pre-VR Knowledge Assessment.
  * User Experience with VR.
  * Effectiveness of Learning.
  * Knowledge Retention and Awareness.
  * Practical Application.
  * Perception of VR as a Learning Tool.
  * Open-Ended Feedback.
  The questionnaire will be administered after participants complete their VR session on pelvic floor anatomy. Responses will be collected electronically to facilitate ease of access and analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Amel Mohamed Yousef, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt